CLINICAL TRIAL: NCT05072574
Title: Assessment of Quality of Life, Nutritional Status and Functional Capacity in People With Advanced Chronic Kidney Disease (CKD) After the Implementation of a Nutritional Education Plan and Individualized Dietary Intervention
Brief Title: Quality of Life, Nutritional Status and Functional Capacity in People With Advanced Chronic Kidney Disease
Acronym: ERCANUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACKD
Record Dates: First submitted 2021-04-08; First posted 2021-10-11 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Diseases
Keywords: Advanced CKD; diet; nutritional education; coaching; quality of life (QoL); nutritional status; functional capacity
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: nutritional education program (Experimental): Specific dietary treatment and follow-up using coaching techniques, supported by new technologies, and will attend a nutritional education program
  Interventions: Other: Specific dietary treatment and follow-up using coaching techniques
- Control Group (No Intervention): Dietary and general lifestyle recommendations

INTERVENTIONS:
Other: Specific dietary treatment and follow-up using coaching techniques — Intervention group will receive specific dietary treatment and follow-up using coaching techniques, supported by new technologies, and will attend a nutritional education program
  Arms: Experimental: nutritional education program

SUMMARY:
This study evaluates the clinical response (quality of life, nutritional status, functional capacity, and disease knowledge) of advanced CKD patients who undergo an individualized dietary intervention and a nutritional education program (group workshops) using motivation coaching techniques, compared to controls who receive general hygiene-nutritional education at every visit.

DETAILED DESCRIPTION:
Randomized study including two parallel groups: patients from the advanced chronic kidney disease (CKD) consulting room of the Malaga University Regional Hospital and controls. The main objective is to assess the clinical response (quality of life, nutritional status, functional capacity, and disease knowledge) of advanced CKD patients who undergo an individualized dietary intervention and a nutritional education program (group workshops) using motivation coaching techniques, compared to controls who receive general hygiene-nutritional education at every visit.

Both groups will be composed of 54 participants. The control group will be provided general dietary and lifestyle recommendations (standard procedure in the nephrology consulting room), whereas the intervention group will receive treatment and individualized dietary follow-up using coaching techniques, supported by information and communication technologies, and will participate in a nutritional education program composed of four on-line sessions.

Two visits (basal and three months after) will be scheduled during the study to obtain and analyse the data. Moreover, in these visits researchers will collect a blood sample in order to perform an assessment of the metabolism, inflammation, and oxidation, and a stool sample in order to evaluate the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

- Patients >18 years old with advanced CKD (GFR <30ml/min) starting follow-up in the advanced CKD consulting room of the Malaga University Regional Hospital and who clearly understand the study and give their informed consent.

Exclusion Criteria:

* Patients presenting any of these conditions:

  * Active cancer
  * Being already participants of another study that may affect the results
  * Pregnancy or possible pregnancy
  * Informed consent refusal
  * Hospital admission during one month previous to the study
  * Severe mental disorders (SMD), prolonged mental disorders involving a high level of disability and social dysfunction, which requires attendance by the mental health and social care network
  * Alcohol or any other substance abuse that, in the researcher's opinion, may interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Assess the clinical response after the quality of life intervention | From baseline to week 12
  Kidney Disease and Quality of Life test (KDQOL-36). The generic component of the KDQOL-36 (items 1-12) is the SF-12, which allows obtaining 2 general scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The specific component of the KDQOL-36 (items 13-36), allows obtaining the scores of the specific subscales for the disease.

SECONDARY OUTCOMES:
Assess the clinical response after intervention in the management of CKD | From baseline to week 12
  Self-Efficacy for Managing Chronic Disease test. The Self-Efficacy Scale for the Management of Chronic Diseases (SEMCD) is made up of 6 items on an analog scale, ranging from 1 (not at all sure) to 10 (totally safe).
  The Spanish version (SEMCD-S) consists of 4 items. A higher number means greater self-efficacy. The scale score is the mean of the items.
Assess the clinical response after the intervention in knowledge about the disease | From baseline to week 12
  Kidney Disease Knowledge Survey test. The Kidney Disease Knowledge Survey (KiKS) instrument consists of 28 items and aims to assess specific knowledge about chronic kidney disease in non-dialysis patients. One point is considered for each correct answer and zero for the incorrect one. The total score is calculated by adding all the correct points and divided by 28, obtaining a value from 0 to 1, with 1 being the highest level of knowledge.
BMI (body mass index) changes | From baseline to week 12
  Measured by body composition analysis
Change in weight | From baseline to week 12
  Weight in kg
Change in fat free body mass | From baseline to week 12
  Fat free body mass in kg assessed by bioelectrical impedance analysis
Change in upper arm circumference | From baseline to week 12
  circumference in cm
Change in arm muscle circumference | From baseline to week 12
  circumference in cm
waist circumference | From baseline to week 12
  circumference in cm
Change in serum potassium concentration (assess kidney function) | From baseline to week 12
  serum potassium in mEq/l
Change in serum phosphorus concentration (assess kidney function) | From baseline to week 12
  serum phosphorus mg/dl
Change in glomerular filtration (assess kidney function) | From baseline to week 12
  Calculated with the formula of CKD-EPI and MDRD and measured in ml/ min/ 1.73 m2
Change in serum albumin concentration | From baseline to week 12
  Serum albumin in g/dl
Change in serum prealbumin concentration | From baseline to week 12
  Serum prealbumin in mg/dl
Change in cholesterol concentration | From baseline to week 12
  Serum cholesterol in mg/dl
Change in HDL concentration | From baseline to week 12
  Serum HDL in mg/dl
Change in LDL concentration | From baseline to week 12
  Serum LDL in mg/dl
Change in TG concentration | From baseline to week 12
  Serum TG in mg/dl
Changes in plasma levels of high sensitivity C reactive protein (hs-CRP) | From baseline to week 12
  Plasma levels of high sensitivity C reactive protein (hs-CRP) in mg/dl
Changes in blood cells | From baseline to week 12
  Blood count
Change in iron concentration | From baseline to week 12
  Serum iron in μg/dl
Change in ferritin concentration | From baseline to week 12
  Serum ferritin in ng/ml
Change in uric acid concentration | From baseline to week 12
  Serum uric acid in mg/dl
Change in urea concentration | From baseline to week 12
  Serum uric acid in mg/dl
Change in magnesium concentration | From baseline to week 12
  Serum magnesium in mg/dl
Change in calcium concentration | From baseline to week 12
  Serum calcium in mg/dl
Change in intact parathyroid hormone (PTHi) concentration | From baseline to week 12
  Serum intact parathyroid hormone (PTHi) in pg/ml
Changes in vitamin D | From baseline to week 12
  Serum vitamin D in ng/ml
Changes in metabolic control | From baseline to week 12
  Measured as HbA1c (glycated hemoglobin)
Assess changes in the degree of depression and / or anxiety | From baseline to week 12
  HADS depression and anxiety symptoms screening test. It is a self-administered scale with 14 items divided into 2 subscales (anxiety and depression) whose maximum score is 21 points for each of them. Based on the score obtained, the patients can be classified as normal (<7), doubtful (between 8 and 10) and potential clinical case (≥ 11). The score is referred to the last week.
Assess the clinical response after the intervention on functional capacity | From baseline to week 12
  Scale of autonomy for activities of daily life "Barthel test". This test measures the capacity of the person to carry out ten basic activities of daily life, obtaining a quantitative estimate of the degree of dependence of the subject. The range of possible IB values is between 0 and 100, with 5-point intervals for the original version. The closer a subject's score is to 0, the more dependency they have; the closer to 100 the more independence.
Assess on functional capacity | From baseline to week 12
  Physical activity test "Short Physical Performance Battery" SPPB. This in turn includes 3 tests: balance, gait speed and getting up and sitting in a chair 5 times. Each test is scored from 0 (worst performance) to 4 (best performance): for the balance test according to a hierarchical combination of performance in the 3 component subtests and for the other 2 tests a score of 0 is assigned to those who do not complete or they attempt the task and scores from 1 to 4 based on the time spent. In addition, a total score for the entire battery is obtained, which is the sum of the 3 tests and ranges from 0 to 12.
Changes on functional capacity: International Physical Activity Questionnaire (IPAQ) | From baseline to week 12
  The International Physical Activity Questionnaire (IPAQ) will be used to evaluate the current physical activity level of the participants. The survey consists of 27 questions and 5 parts.
Change from Handgrip Strength | From baseline to week 12
  Strength will be recorded by Jamar Hydraulic Hand Dynamometer (Kg)
Characterize exercise participant behavior | From baseline to week 12
  International Physical Activity Questionnaire (IPAQ). The IPAQ consists of 7 questions about the frequency, duration and intensity of activity (moderate and intense) carried out in the last seven days, as well as walking and sitting time in a work day. It evaluates three characteristics of physics (PA): intensity (mild, moderate or vigorous), frequency (days per week) and duration (time per day). Weekly activity is recorded in Mets (Metabolic Equivalent of Task or Metabolic Index Units) per minute and week.
Change in handgrip strength | From baseline to week 12
  Handgrip strength in kg, measured by the jamar hydraulic hand dynamometer.
Changes the clinical response after the intervention in blood pressure figures (mmHg). | From baseline to week 12
  Assess if syastolic and diastolic pressure improves after training and at 6 months of follow-up.
Diet composition: PREDIMED test (Prevention with Mediterranean Diet) | From baseline to week 12
  Adherence to the Predimed Plus diet pattern 17 (0 - minimum adherence, 17 - maximum adherence)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Olveira, MD, PhD, Principal Investigator — Hospital Regional Universitario de Málaga - FIMABIS
Locations (1):
- Hospital Regional Universitario de Málaga, Málaga, Spain

REFERENCES:
- [Derived] Padial M, Rebollo A, Jimenez-Salcedo T, Lopez V, Avesani CM, Lindholm B, Qureshi AR, Olveira G. A Pilot Clinical Trial of a Nutrition Education Program on Quality of Life in CKD. Clin J Am Soc Nephrol. 2025 Oct 1;20(10):1352-1364. doi: 10.2215/CJN.0000000790. Epub 2025 Aug 19. PMID 40828609